CLINICAL TRIAL: NCT03629457
Title: Efficacy of a Training Program in Mindfulness and Self-Compassion of 4 Sessions in Front of the 8 Sessions to Reduce Work Stress and Burnout in Professionals of Medicine and Nursing (MINDUUDD Project)
Brief Title: Efficacy of a Mindfulness Program to Reduce Stress and Burnout in Professionals of Medicine and Nursing (MINDUUDD)
Acronym: MINDUUDD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luis A Perula (Other Government)
Collaborators: Sociedad Andaluza de Medicina Familiar y Comunitaria (Unknown)
Responsible Party: Sponsor-Investigator, Luis A Perula, Doctor in medicine. Specialist in Preventive Medicine and Public Health. Health Technician Teaching Unit Family and Community Medicine, Hospital Universitario Reina Sofia de Cordoba
Organization: Hospital Universitario Reina Sofia de Cordoba (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MINDUUDD
Record Dates: First submitted 2018-08-02; First posted 2018-08-14 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Stress; Burnout Syndrome
MeSH Terms: conditions — Burnout, Psychological | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group 4s (mindfulness) (Experimental): Abbreviated program of 4 weeks: will consist of 4 weekly sessions of 2 hours. Participants must practice at home for 15 minutes a day
  Interventions: Behavioral: Mindfulness and Mindful Self-Compassion
- Intervention group 8s (mindfulness) (Experimental): Program of 8 weeks: The format will be 8 weekly sessions of 2 hours. Participants must practice at home for 30 minutes a day
  Interventions: Behavioral: Mindfulness and Mindful Self-Compassion
- Control group (No Intervention): The participants will only receive a one-hour information session and will be invited to complete the questionnaires provided in two moments of the time (coinciding with the interventions in the experimental groups)

INTERVENTIONS:
Behavioral: Mindfulness and Mindful Self-Compassion — Mindfulness Based Stress Reduction (MBSR) and Mindful Self-Compassion
  Arms: Intervention group 4s (mindfulness); Intervention group 8s (mindfulness)

SUMMARY:
The objective is to check whether a training program in mindfulness and self-pity based on a 4-session intervention (abbreviated program) is as effective as the standard 8-session MBSR program in reducing work stress and burnout in tutors and residents of Medicine and Family and Community Nursing.

It is a controlled clinical trial, randomized by cluster, of three parallel arms, multicentric. Six teaching units (ratio 1: 1: 1) will be randomized to one of the three study groups: 1) Experimental Group-8 (EG8); 2) Experimental Group-4 (EG4); 3) Control group (CG).

At least 132 subjects will participate, 44 in the EG8, 44 in the EG4 and 44 in the CG.

The interventions will be based on the MBSR (Mindfulness Based Stress Reduction) program, to which some of the practices of the MSC (Mindful Self-Compassion) program will be added.

The EG8 intervention will be carried out during 8 weekly sessions of 2.5 hours, while the EG4 intervention will be of 4 sessions of 2.5 hours. The participants will have to practice at home for 30 minutes / day in the EG8 and 15 minutes / day in the EG4.

In the 3 groups the questionnaires FFMQ (mindfulness), SCS (self-pity), ordinal scale (0-10) and questionnaire PSQ (perceived stress) and MBI (burnout) will be passed. Empathy will also be measured, through the EEMJ, anxiety and depression disorders (EADG) and self-perceived health status.

ELIGIBILITY:
Inclusion Criteria:

* Health professionals (doctors and nurses tutors and residents) assigned to 6 teaching units of family and community care, which are active.

Exclusion Criteria:

* That you have previously done a training course or workshop in mindfulness of at least 4 weeks.
* That during the field work they are in a situation of prolonged or long-term sick leave.
* Have mental disorders that discourage the intervention.
* That they do not give their informed consent to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Degree of occupational stress | Change from baseline at 4 weeks (EG4) or 8 weeks (EG8 or CG)
  An ordinal scale that ranges from 0 (no degree of stress) to 10 (maximum degree of stress) stress, will be used
Degree of occupational stress | Change from baseline at 4 weeks (EG4) or 8 weeks (EG8 or CG)
  PSQ questionnaire (Perceived Stress Questionnaire). It consists of 30 items that can be scored using a Likert scale (1 to 4). Higher total values indicate more stress.
Degree of burnout | Change from baseline at 4 weeks (EG4) or 8 weeks (EG8 or CG)
  Maslach Burnout Inventory-General Survey (MBI). Spanish version of the MBI-HSS25. It consists of 22 scoring items from 0 to 6 that measure the three dimensions of the syndrome: emotional fatigue (CE), 9 items and a maximum score of 54 points; depersonalization (DP), 5 items and maximum score of 30 points; personal fulfillment (RP), 8 items and maximum score of 48 points. The cut points used were: emotional fatigue under <19, moderate 19-26, high> 26. Depersonalization under <6, moderate 6-9, high> 9. Personal performance under> 39, moderate 39-34, high <34 .
Degree of Self-Compassion | Change from baseline at 4 weeks (EG4) or 8 weeks (EG8 or CG)
  Self-compassion questionnaire. The short scale of the Spanish version, validated by García-Campayo et al, will be used, with 12 items scored using a Likert scale (1 to 5) that measures how the subject usually acts towards himself in difficult moments. It consists of six subscales: self-friendliness, common humanity, mindfulness, and their opposites: self-judgment, isolation and over-identification. Higher total values indicate more self-pity.

SECONDARY OUTCOMES:
Degree of empathy | Change from baseline at 4 weeks (EG4) or 8 weeks (EG8 or CG)
  Jefferson Medical Empathy Scale (EEMJ), HP version. Defines empathy based on three factors: "perspective taking", "compassionate care" and the ability to "put yourself in the patient's shoes". It has a minimum score of 20, maximum of 140 and does not establish a cut-off point, it contains 20 Likert-type items on a 7-point scale. There are 10 items written in the positive sense and 10 in the negative sense.

OTHER OUTCOMES:
Anxiety and Depression | Change from baseline at 4 weeks (EG4) or 8 weeks (EG8 or CG)
  Goldberg Anxiety and Depression Scale (GADS, EADG in spanish versión). It consists of two sub-scales, one of anxiety and the other of depression. Each sub-scale has 9 items of dichotomous response (Yes / No) and are structured in 4 initial items of screening, to determine whether or not there is likely to be a mental disorder, and a second group of 5 items that are formulated if you get positive answers to the screening questions (2 or more for anxiety and more than 1 for depression), but in the investigation the full scale is usually applied, and that way it was used in the present study. an independent score for each scale, with a point for each affirmative answer. Goldberg et al have proposed cutoff points ≥ 4 for the anxiety scale, and ≥ 2 for depression.
Self-perceived health status | Change from baseline at 4 weeks (EG4) or 8 weeks (EG8 or CG)
  Ordinal cualitativ scale: Very bad, bad, good or excellent

CONTACTS AND LOCATIONS:
Locations (1):
- Family Medicine Teaching Unit and Community, Córdoba, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Magallon-Botaya R, Perula-de Torres LA, Verdes-Montenegro Atalaya JC, Perula-Jimenez C, Lietor-Villajos N, Bartolome-Moreno C, Garcia-Campayo J, Moreno-Martos H; Minduudd Collaborative Study Group. Mindfulness in primary care healthcare and teaching professionals and its relationship with stress at work: a multicentric cross-sectional study. BMC Fam Pract. 2021 Feb 2;22(1):29. doi: 10.1186/s12875-021-01375-2. PMID 33530929
- [Derived] Perula-de Torres LA, Atalaya JCV, Garcia-Campayo J, Roldan-Villalobos A, Magallon-Botaya R, Bartolome-Moreno C, Moreno-Martos H, Melus-Palazon E, Lietor-Villajos N, Valverde-Bolivar FJ, Hachem-Salas N, Rodriguez LA, Navarro-Gil M, Epstein R, Cabezon-Crespo A, Moreno CM; collaborative group of the MINDUUDD study. Controlled clinical trial comparing the effectiveness of a mindfulness and self-compassion 4-session programme versus an 8-session programme to reduce work stress and burnout in family and community medicine physicians and nurses: MINDUUDD study protocol. BMC Fam Pract. 2019 Feb 6;20(1):24. doi: 10.1186/s12875-019-0913-z. PMID 30727962